CLINICAL TRIAL: NCT05344651
Title: Comparing the Baerveldt and Paul Glaucoma Drainage Devices and Their Effects on the Corneal Endothelium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oogziekenhuis Rotterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OZR-2020-30; NL80518.078.22 (Other: Centrale Commissie Mensgebonden Onderzoek); MEC-2022-0069 (Other: Medical Ethical Committe of the Erasmus Medical Center)
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baerveldt glaucoma drainage device (Active Comparator)
  Interventions: Device: Surgery/implantation
- Paul glaucoma drainage device (Experimental)
  Interventions: Device: Surgery/implantation

INTERVENTIONS:
Device: Surgery/implantation — The glaucoma drainage device consists of a plate and a tube. During surgery the plate is positioned underneath the conjunctiva and two extraocular muscles in the upper temporal quadrant of the eye. The tube is positioned in the anterior chamber.

SUMMARY:
Rationale: The Baerveldt glaucoma drainage device (GDD) successfully reduces intraocular pressure but also involves a risk of corneal endothelial deterioration. Supposedly, the tip of a GDD tube with a thinner diameter, such as the Paul implant, will remain at a larger distance from the cornea and, thereby, cause less damage.

Objective: To determine whether the Paul tube induces less damage to the corneal endothelium than the Baerveldt GDD.

Study design: Randomized clinical trial. Study population: Phakic patients scheduled for surgical GDD implantation. Intervention: Either a Baerveldt or a Paul GDD implant. Main study parameters/endpoints: Endothelial cell density and tube position at 24 months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The Paul GDD may have a less harmful effect on corneal endothelium. Otherwise, both GDDs will probably have a similar risk/benefit profile. The risks of study-related assessments are negligible, burden is low, extra time is about 5 x 1.5 h (total 7.5 h) in two years.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Informed consent.
* Caucasian ethnicity (to facilitate comparison of results with those of earlier work). Ethnicity will be based on self-reported origin of subject and/or parents.
* Primary open-angle glaucoma, pseudoexfoliative glaucoma, or pigmentary glaucoma.

Exclusion Criteria:

* History of intraocular surgery (e.g. vitrectomy, cataract surgery, cyclodestructive procedures etc).
* History of ocular comorbidity (e.g. active uveitis, proliferative diabetic retinopathy).
* Pseudophakia.
* Functionally monocular patients.
* Need for glaucoma surgery combined with other ocular procedures (i.e. cataract surgery, keratoplasty, or retinal surgery) or an anticipated need for additional ocular surgery.
* Narrow anterior chamber angle.
* Best corrected visual acuity less than 0.1.
* Severe blepharitis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change of endothelial cell density (ECD). | Baseline and 2 years
  ECD will be assessed at the center of the cornea and close to the tube.

SECONDARY OUTCOMES:
Endothelial cell density (ECD). | Baseline, 3, 6, 12, 24 months.
  ECD will be assessed at the center of the cornea and close to the tube.
Intraocular pressure. | Baseline, 1, 3, 6, 12, 24 months.
  Intraocular pressure.
Orthoptic assessment. | Baseline, 3, 6, 12, 24 months.
  Prism cover test: total deviation at 30 cm; Goldmann: monocular ductions in 8 directions starting from primary position, binocular field of single vision.

CONTACTS AND LOCATIONS:
Locations (1):
- Oogziekenhuis Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No